CLINICAL TRIAL: NCT02399592
Title: Tocotrienol as a Nutritional Supplement in Patients With Advanced Ovarian Cancer
Acronym: Toco-Ovar
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Toco-Ovar
Record Dates: First submitted 2015-03-20; First posted 2015-03-26 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-02

CONDITIONS: Ovarian Cancer
Keywords: Platinum resistant
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab and Tocotrienol (Experimental)
  Interventions: Drug: Bevacizumab; Drug: Tocotrinol

INTERVENTIONS:
Drug: Bevacizumab — 10 mg/kg q3w
Drug: Tocotrinol — 300 mg tid

SUMMARY:
The purpose of this study is to to investigate the effect of tocotrienol as a nutritional supplement in combination with bevacizumab in patients with advanced ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed epithelial, primary fallopian or primary peritoneal cancer.
* Prior treatment with at least two different cytostatic regimens including platinum.
* Progression on previous treatment.
* Measurable disease by RECIST 1.1 or evaluable by GCIG CA-125 criteria.
* Age ≥ 18 years.
* Performance stage 0-2.
* Adequate bone marrow function, liver function, and renal function (within 7 days prior to inclusion):

  * WBC ≥ 3.0 * 10^9/l or neutrophils (ANC) ≥ 1.5 * 109/l
  * Platelet count ≥ 100 * 10^9/l
  * Hemoglobin ≥ 6 mmol/l
  * Serum bilirubin < 2.0 * ULN
  * Serum transaminase ≤ 2.5 * ULN
  * Serum creatinine ≤ 1.5 ULN
* Urine dipstick for protein <2+. If the dipstick shows protein ≥2+ 24 hour urine testing must be made with protein contents < 1 g.
* Written informed consent.

Exclusion Criteria:

* Other malignant diseases within 5 years prior to inclusion in the study, except curatively treated basal cell or squamous cell carcinoma of the skin and other types of cancer with minimal risk of recurrence.
* Other experimental therapy or participation in another clinical trial within 28 days prior to treatment initiation.
* Underlying medical disease not adequately treated (diabetes, cardiac disease).
* Uncontrolled hypertension (BT >150/100 despite antihypertensive treatment).
* Surgery, incl. open biopsy, within 4 weeks prior to first dose of bevacizumab.
* Non-healing wounds or fractures.
* Cerebral vascular attack, transient ischemic attack or subarachnoidal hemorhage within 6 months before start of treatment.
* Clinically significant cardiovascular disease, including:

  * Myocardial infarction or unstable angina within 6 months before start of treatment
  * New York heart Association (NYHA) class ≥ 2
  * Poorly controlled cardiac arrhythmia despite medication
  * Periferal vascular disease grade ≥ 3
* Allergy to the active substance or any of the auxiliary agents
* Bleeding tumor
* Pregnant or breast-feeding patients. For fertile women a negative pregnancy test at screening is mandatory.
* Fertile patients not willing to use effective methods of contraception during treatment and for 6 months after the end of treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Fraction of patients without progression after six months of treatment | 6 months after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anders Jakobsen, DMSc, Study Chair — Department of Oncology, Vejle Hospital
Locations (1):
- Department of Oncology, Vejle Hospital, Vejle, Denmark